CLINICAL TRIAL: NCT07149103
Title: A Pilot Sham-Controlled Study to Evaluate the Safety and Efficacy of a Wearable Microneedle Percutaneous Neuromodulation System for Idiopathic Overactive Bladder and Urinary Incontinence
Brief Title: Stimulating Percutaneous Array for Urinary Reflex Control (SPARC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australis Scientific PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-001
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Over Active Bladder
Keywords: Over active bladder; Incontinence; Ideopathic Over active bladder; Percutaneous Tibial Nerve Stimulation (PTNS)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): The treatment arm will undergo the experimental treatment
  Interventions: Other: Percutaneous Tibial Nerve Stimulation
- SHAM ARM (Placebo Comparator): The sham arm will undergo the same procedure as the treatment group but the therapy will not be switched on
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Percutaneous Tibial Nerve Stimulation — By wearing the Confidanz Smart Patch, the Tibial Nerve will be stimulated
  Arms: Treatment Arm
Other: Placebo — No active stimulation will be provided
  Arms: SHAM ARM

SUMMARY:
The Confidanz Smart Patch System consists of a Smart Patch containing one transcutaneous gel electrode and one percutaneous microneedle array electrode that sits directly superficial to the posterior tibial nerve. An applicator is used by the patient to deploy the microneedles into the skin. A Capital Stimulation Unit (CSU) is magnetically aligned with the Smart Patch and generates biphasic current wave form to the posterior tibial nerve through the patch. The CSU is connected to a mobile application via Bluetooth, allowing control over the stimulation intensity parameters.

Primary Objective: To investigate the safety of the Confidanz Smart Patch System for adults diagnosed with idiopathic overactive bladder.

Secondary Objective: To measure the reduction from baseline in average incontinence events (IE) per day at 6- and 12-weeks.

Primary Hypothesis: The use of the Confidanz Smart Patch System is safe for use in adults with idiopathic overactive bladder.

DETAILED DESCRIPTION:
The Clinical Trial is a Randomised, single-blinded, sham-controlled study designed to assess the safety and performance of the Confidanz Smart Patch System for home-based intermittent use under clinical supervision, in patients with overactive bladder systems. Participant screening will occur at least 3-days prior to the baseline visit in the clinic. Participants who meet all the inclusion criteria and none of the exclusion criteria will be enrolled. Up to 40 participants will be enrolled in this clinical investigation. A computer-generated sequence will be created using a block randomisation method, participants will be randomised in a 3:1 fashion.

At the baseline visit, the investigator or study staff member will train the participant on the correct use of the device. At-home weekly treatments will be conducted for 12 weeks, here the patient will apply the Smart Patch and initiate a 30-minute stimulation session through the mobile application. The treatment arm will receive stimulation, whereas the control arm will not. Symptom tracking and adverse events will be recorded.

A maximum total of 12 weekly treatments will be conducted. At baseline, 6 and 12 weeks, a 3-day bladder diary, International Consultation on Incontinence Questionnaire (ICIQ), the Overactive Bladder Symptom Score (OABSS), Short Form Survey SF-12, Patient Global Impression of Change (PGI-C), VAS pain scale, and participant decision-making and feedback questionnaire will be administered in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent for participation in the investigation
2. Is aged 18 years or older
3. Has been diagnosed with idiopathic overactive bladder (OAB) by a qualified urologist (FRACS) or gynaecologist (FRANZCOG)
4. Eligibility is based on meeting the criteria for an OAB, defined by the International Continence Society as an average urinary frequency: ≥8 voids and ≥1 urgency episode (with or without incontinence) per 24 hours
5. Clinically acceptable laboratory results within 30 days of enrolment Urinalysis: Dipstick (Leukocytes & Nitrites)
6. In the Investigator's opinion, participant is able and willing to comply with all trial requirements
7. Willing to allow their general practitioner and/or other specialists to be aware of their participation in the trial.

Exclusion Criteria:

1. Presence of urinary tract infection based on a positive dipstick AND positive mid-stream urine (MSU) test within 4 weeks prior to therapy commencement.
2. Female participant who is pregnant, lactating or planning pregnancy during the trial.
3. History of bladder augmentation/cystoplasty
4. Morbid obesity (BMI greater than 35)
5. Poorly controlled diabetes mellitus (HbA1c > 7.5% (based on diabetic study)
6. Intravesical injection of botulinum toxin within 12 months of study enrolment.
7. Patients who have failed intravesical Botox therapy.
8. Patients with neurogenic lower urinary tract dysfunction or relevant neurological disease
9. A treatment within the previous year of neuromodulation (TNS or sacral neuromodulation) for OAB.
10. Participant with pacemakers or implantable defibrillators, or other active implantable devices (e.g., spinal cord stimulators, bladder neurostimulators)
11. Participant who have participated in another research trial involving an investigational product in the past 12 weeks.
12. Participant on medication therapy for OAB who have not gone through a two-week washout period during which time medications were discontinued.
13. Participant is in the investigators opinion, unable to comply with trial requirements.
14. Participant has inflamed, infected or otherwise compromised skin in the treatment area.
15. Participant with a bleeding disorder e.g., haemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 12 weeks
  Number of AEs and SAEs occurring throughout the study

SECONDARY OUTCOMES:
Change from baseline in average voids per day at 6- and 12-weeks. | Up to 12 weeks
  To measure and compare average incontinence events (IE) per day at 6- and 12-weeks from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Vincent Tse Pty Ltd, Chatswood, New South Wales
  - AndroUrology Centre, Spring Hill, Queensland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.